CLINICAL TRIAL: NCT06138860
Title: Effect of Strain Counter Strain Technique in Treatment of Lower Back Myofascial Pain Syndrome: a Randomized Controlled Clinical Trial
Brief Title: Effect of Strain Counter Strain Technique in Treatment of Lower Back Myofascial Pain Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Collaborators: King Khalid University (Other)
Responsible Party: Principal Investigator, Doaa Ayoub Elimy Mohammed, Lecturer of physical therapy for basic science department., faculty of physical Therapy, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ECM#2023-1101; HAPO-06-B-001
Record Dates: First submitted 2023-11-11; First posted 2023-11-18 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-03

CONDITIONS: Lower Back Myofascial Pain Syndrome
Keywords: Low back Pain; Myofascial pain syndrome; Strain counter strain technique; trigger point
MeSH Terms: conditions — Low Back Pain; Myofascial Pain Syndromes | interventions — Exercise Therapy

STUDY DESIGN:
Intervention Model Description: strain counter strain technique and physical therapy exercises
Who Masked: Investigator, Outcomes Assessor
Masking Description: random generator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- strain counter strain technique (Experimental): the patients will receive strain counter strain technique plus physical therapy exercises three times a week for four weeks
  Interventions: Other: strain counter strain technique; Other: physical therapy exercises
- physical therapy exercises (Active Comparator): the patients will receive physical therapy exercise three times a week for four week
  Interventions: Other: physical therapy exercises

INTERVENTIONS:
Other: strain counter strain technique — It will be done in accordance with the technique principles in which the therapist will locate trigger point, and then find a position of comfort or mobile point (at least a 70% decrease in tenderness),monitored the tender point, holding the position o f comfort for 90 seconds, It will be conducted three times per session, for twelve sessions three times per week every other day over the course of a month.
  Arms: strain counter strain technique
Other: physical therapy exercises — Physical therapy exercises for twelve sessions, three times a week, over the course of a month.
  Exercises will include:
  stretching exercises for the hamstring, calf muscles, and back muscles.
  strengthening exercises for back muscles and abdominal muscles.

SUMMARY:
This study aims to investigate the impact of impact of strain counterstrain technique on pain, lumbar range of motion and functional impairment in patients with lower back Myofascial pain syndrome.

DETAILED DESCRIPTION:
Myofascial Pain Syndrome (MPS) is a prevalent form of musculoskeletal pain that impedes everyday activities and reduces productivity.Those who experience difficulties with regional pain frequently report myofascial pain. According to statistics, between 85% and 93% of patients who attend specialized pain treatment facilities and between 21% and 30% of people with regional pain who visit a general medical clinic also have it.Trigger points, which are hyperirritable tender spots in palpably tense bands of skeletal muscles, are what define it. These spots can cause referred pain patterns, painfully limited range of motion, stiffness, muscle fatigue, and autonomic dysfunction.

Numerous clinical therapies as well as training regimens have been developed to combat trigger points. Strain counterstrain technique (SCS), is one of several manual methods for trigger points, which is a passive method that opens shortened tissues and reduces musculoskeletal pain. It may be possible to activate the Golgi tendon organ, which relaxes tense and tight muscles, by positioning shortened and painful tissues in a comfortable way, which would result in a reduction in the sensitivity of the trigger point.

Hence, the purpose of this study is to ascertain how SCS affects pain, ROM, and functional disability in individuals suffering from lower back myofascial pain syndrome.

ELIGIBILITY:
Inclusion Criteria:

1. The patients age from 20 to 40 years for both genders.
2. Patients (office worker) with mechanical back pain for 3 months ago and has not been diagnose as a specific disease or spinal abnormality.
3. Patients suffering from active MTrPS in lower back muscle.
4. According to the Oswestry Low Back Pain Disability Questionnaire, patients suffered moderate disability care (20-40%).
5. Patients capable of doing ROM assessment of Lumbar Spine (flexion, extension, as well as side binding) within the limit of pain.

Exclusion Criteria:

1. Neurological, systemic illness and infectious diseases such as rheumatologic diseases, tumor.
2. Psychiatric/mental deficit.
3. Patients who had a previous surgical history (within 6 months) were also excluded prior to the baseline assessment.
4. Vertebral compression fracture
5. Pregnancy and lactation.
6. Existing lower limb symptoms.
7. Activity intolerance due to cardiopulmonary disease.

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-02-29 (Actual); Study Completion 2024-02-29 (Actual)

PRIMARY OUTCOMES:
pain intensity | up to four weeks
  A Visual Analogue Scale (VAS) will be used by the patient to mark his or her level of pain, usually 10 cm long, ranging from no pain or discomfort (zero) to the worst pain that the patient can possibly feel.

SECONDARY OUTCOMES:
range of motion assessment | up to four weeks
  inclinometer will be used to assess lumbar flexion, extension and side bending
functional impairment | up to four weeks
  Arabic version of Oswestry Disability Index will be used for assessment of functional disability

CONTACTS AND LOCATIONS:
Overall Officials: Ghada MR Koura, Ass. prof, Study Director — King Khalid University, Saudi Arabia
Locations (1):
- Ghada Mohamed Rashad Koura, Abhā, Saudi Arabia